CLINICAL TRIAL: NCT04914650
Title: TEleRehabilitation Nepal (TERN) to Improve Quality of Life of People With Spinal Cord Injury and Acquired Brain Injury. A Proof-of-concept Study
Brief Title: TEleRehabilitation Nepal (TERN) to Improve Quality of Life of People With Spinal Cord Injury and Acquired Brain Injury
Acronym: TERN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Spinal Injury Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Dr Manoj Sivan, Dr, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MREC 19-031
Record Dates: First submitted 2021-06-03; First posted 2021-06-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injuries; Traumatic Brain Injury; Acquired Brain Injury, Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries, Traumatic; Brain Injuries; Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation intervention (Experimental)
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Providing multidisciplinary rehabilitation to individuals with spinal cord injury or brain injury using virtual conference methods

SUMMARY:
Nepal is a low-income country with over 3 million individuals with physical disabilities and currently no government-run specialist rehabilitation services. The aim of this research proposal is to work in partnership with a Nepal Non-Governmental Organisation (NGO), the Spinal Injury Rehabilitation Centre (SIRC, Nepal) to achieve the following:

1. estimate the rehabilitation needs in individuals after stroke, brain injury and spinal cord injury in rural communities after discharge from SIRC
2. hold user and stakeholder workshops to explore the role of multidisciplinary teleconferencing methods for remote assessment and management and agree systems for piloting
3. deploy and pilot a novel telerehabilitation system to improve the lives of these individuals, and evaluate it in terms of feasibility and acceptability

DETAILED DESCRIPTION:
The methods to be used in each of the three work packages of this study are:

Work Package 1: Identifying baseline and context

Individuals discharged from SIRC between January 2018 and December 2019 will be identified and recruited to the study. Initially, a cross sectional study will capture their experiences and baseline community outcomes using both standardised quantitative outcome measures and qualitative data from semi-structured interviews. Recruitment and data collection for this part of the study will be conducted by partners in Nepal. Analysis and management of this data will be joint between Nepal and Leeds teams.

Work Package 2: Assessing utility of telerehabilitation to address needs

Informed by previous work package, user and stakeholder workshops will be used to explore the role of multidisciplinary video teleconferencing, telemedicine follow-up clinics, remote management using mobile phone camera monitoring and other methods identified to reach consensus on interventions to address the most pressing clinical challenges. These workshops will be facilitated by all the researchers and will involve service users, family members, clinicians, hospital managers, community health providers, NGO representatives and national policy makers.

Work Package 3: Pilot and rapid evaluation

The telerehabilitation interventions agreed in work package 2 will then be piloted by the clinical team at SIRC and the participants recruited in work package 1. This will involve post discharge follow up facilitated by the telerehabilitation system, and may result in further clinical rehabilitation care as appropriate (advice, provision of equipment, etc.).

This is followed by a rapid, mixed-methods evaluation which will assess of the feasibility and acceptability of telerehabilitation interventions by incorporating:

* analysis of routinely collected clinical caseload data
* standardised quantitative outcome measures
* semi-structured interviews with service user participants and focus group discussions with staff
* case studies of exemplar cases including video recording

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or above Diagnosis of spinal cord injury or acquired brain injury and received inpatient care in SIRC Discharged from SIRC between February 2018 and August 2019.

Exclusion Criteria:

Individuals who do not report any ongoing rehabilitation needs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | 6 months
  Modified Barthel Index

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale | 6 months
  Depression Anxiety Stress Scale
EuroQoL | 6 months
  EuroQoL

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sivan, MD, Principal Investigator — University of Leeds
Locations (1):
- Spinal Injury Rehabilitation Centre, Bhainsepati, Kavre, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhakal R, Baniya M, Solomon RM, Rana C, Ghimire P, Hariharan R, Makower SG, Meng W, Halpin S, Xie SQ, O'Connor RJ, Allsop MJ, Sivan M. TEleRehabilitation Nepal (TERN) for People With Spinal Cord Injury and Acquired Brain Injury: A Feasibility Study. Rehabil Process Outcome. 2022 Oct 18;11:11795727221126070. doi: 10.1177/11795727221126070. eCollection 2022. PMID 36278119